CLINICAL TRIAL: NCT04935073
Title: A Randomized Controlled Study on the Short-term Intervention of Traditional Chinese Medicine Herbs in the Freeze-all IVF Cycle to Improve Pregnancy Rate
Brief Title: Traditional Chinese Medicine Herbs in the Freeze-all IVF Cycle
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-M2020442
Record Dates: First submitted 2021-05-13; First posted 2021-06-22 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Infertility, Female
Keywords: infertility; traditional chinese medicine; freeze-all IVF cycle; Embryo Transfer
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — si-wu-tang; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine herbs treatment group (Experimental): the treatment group will receive treatment with the Chinese herbal formula on the 5th day of the menstrual cycle and lasts to 14 days after IVF-ET.
  Interventions: Drug: Prescription of traditional Chinese Medicine named Er Zhi Wan combined with Si Wu Tang; Drug: Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection
- Western medicine group (Active Comparator): The control group will be treated with conventional Western medicine
  Interventions: Drug: Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection

INTERVENTIONS:
Drug: Prescription of traditional Chinese Medicine named Er Zhi Wan combined with Si Wu Tang — The medicines used in this study including Radix et Rhizoma Ligustrum 15 g, Radix Morindae Sinensis 12 g, Fructus Lycii 15 g, Semen Cuscutae 20 g, Radix Rehmanniae 15 g, Radix Angelicae Sinensis 10 g, Radix Paeoniae Alba 10 g, Ligusticum wallichii 6 g, Poria cocos 15g, Polygonatum 15g, eclipta 10g. which will be taken for 10-15days.After the ET, the treatment group will continue to take Chinese herbal medicine, changing to Shou Tai pills ( Morinda officinalis 15 g, Teasel 15g，Cuscutae 20 g, Eucommia ulmoides 15 g, Rehmannia 15 g, Cornus officinalis 15 g, loranthus parasiticus 20 g, Ligustrum lucidum 15g, Salvia miltiorrhiza 10g, Scutellaria baicalensis 10g, Atractylodes macrocephala 15g); which will be taken for 14days. The hospital will be responsible for the decoction of 200 mL per dose, 1 dose per day, divided into 2 doses in the morning and in the evening.
  Other Names: conventional western medicine(Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection )
  Arms: Traditional Chinese Medicine herbs treatment group
Drug: Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection — The intervention starts from the 5th day of the menstrual cycle and lasts to the day before IVF-ET.

SUMMARY:
In the early stage, the preliminary study found that traditional Chinese medicine (TCM) intervention aimed at Nourishing kidney and regulating blood circulation in freeze-all IVF cycles can improve the clinical pregnancy rate. In order to further study the role of TCM in improving the pregnancy outcome of IVF-ET in infertility. A randomized controlled clinical trial will be used in this study. 90 infertile patients are randomly divided into two groups. The control group will be treated with conventional modern medicine, and the treatment group will be treated with traditional Chinese herbs on the basis of conventional modern medicine. The intervention starts from the 5th day of the menstrual cycle and lasts until the day before IVF-ET. After the transplantation, the TCM treatment continues for 14 days. The number of oocytes, antral follicles, AMH, serum FSH, and clinical pregnancy rate will be observed to evaluate the effect of TCM herbs on the improvement of pregnancy outcomes. In addition, all the participants will be asked to complete the self-evaluation of the anxiety/depression scale on the 7th day of the menstrual cycle, before and after transplantation, to analyze the emotional changes of the subjects during the study. The study will also observe the safety and health economic indicators of TCM treatment, so as to improve the overall efficacy of TCM Combined Application in assisted reproductive technology in the future.

DETAILED DESCRIPTION:
The trial is designed as a randomized, controlled clinical trial with two groups established by 1:1 equal allocation, a treatment group with interventions using herbs to tonify the kidneys and regulate blood and a control group treated using conventional Western medicine. Random numbers will be prepared by an independent third-party statistician who prepared a list of random group codes for this study. Enrolled subjects will be given a subject number during the screening process and, upon formal enrolment, will be randomly assigned to either the test or control group with a corresponding random number.

Interventions Treatment method Phase 1: The control group will be treated with conventional Western medicine, whereas the treatment group will receive treatment with the Chinese herbal formula. Treatment with the Chinese herbal formula will start on the 5th day of menstruation cycle. The medicines used will be Er Zhi Wan combined with Si Wu Tang (Radix et Rhizoma Ligustrum 15 g, Radix Morindae Sinensis 12 g, Fructus Lycii 15 g, Semen Cuscutae 20 g, Radix Rehmanniae 15 g, Radix Angelicae Sinensis 10 g, Radix Paeoniae Alba 10 g, Ligusticum wallichii 6 g, Poria cocos 15g,Polygonatum 15g,eclipta 10g); which will be taken for 10-15days.

Phase 2: After ET, the control group will be treated conventionally with no TCM intervention, and the treatment group will continue to take Chinese herbal medicine, changing to Shou Tai pills ( Morinda officinalis 15 g, Teasel 15g，Cuscutae 20 g, Eucommia ulmoides 15 g, Rehmannia 15 g, Cornus officinalis 15 g, loranthus parasiticus 20 g, Ligustrum lucidum 15g, Salvia miltiorrhiza 10g, Scutellaria baicalensis 10g, Atractylodes macrocephala 15g); which will be taken for 14days. The hospital will be responsible for the decoction of 200 mL per dose, 1 dose per day, divided into 2 doses in the morning and in the evening.

Serum human chorionic gonadotropin (hCG) will be measured, and an hCG>30 IU will be considered to indicate biochemical pregnancy. Ultrasound monitoring will be performed 30 days after ET to calculate the clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for infertility.
2. Meet the criteria for identifying kidney deficiency in TCM.
3. Patients who Planning to undergo IVF-ET for pregnancy in our center, Age ≤40 years and ≥25 years.
4. Previous embryo transfer failure ≥ 2 times.
5. Menstrual cycle is basically normal, and normal ovulation has been monitored in the past.
6. There were more than 1 blastocyst /more than 2 high-quality embryos with more than 6 cells on day 3/more than 2 high-quality embryos with more than 4 cells on day 2.
7. Consent to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Patients with endometritis, acute pelvic inflammatory disease, mycotic vaginitis, bacterial vaginitis, adnexitis or other systemic infections.
2. It has been confirmed that there are obvious and serious other organic lesions in the reproductive organs.
3. Patients with allergic constitution
4. Infertility caused by genetic factors
5. Patients with serious primary diseases such as cardio cerebrovascular, kidney, liver and hematopoietic system and psychosis
6. A person who is unable to cooperate (such as a combination of neurological or mental illness, or a reluctance to cooperate)
7. The endometrial thickness on the day of hCG was less than 6 mm or the endometrial morphology on the day of hCG was type C
8. Those who did not agree to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate (%) | up to 6 weeks from enrollment
  Follow up by telephone calls 14days after the IVF-ET

SECONDARY OUTCOMES:
Concentration of β-human Choriogonadotropin(β-HCG) | up to 6 weeks from enrollment
  Obtained by blood sampling 14days after the proposed IVF-ET

OTHER OUTCOMES:
Changes from Baseline concentration of Self rating Anxiety Scale (SAS) | The 5th day of menstruation、 immediately before the proposed IVF-ET procedure、14 days after the IVF-ET
  They were completed on the 5th day of menstruation, before transplantation and the 14th day after transplantation.If the total score of anxiety is less than 50, it is normal; 50-60 was mild, 61-70 was moderate, and over 70 was severe anxiety
Changes from Baseline concentration of Self rating Depression Scale (SDS) | The 5th day of menstruation、 immediately before the proposed IVF-ET procedure、14 days after the IVF-ET
  They were completed on the 5th day of menstruation, before transplantation and the 14th day after transplantation.Under normal circumstances，the maximum values of SDS gross score is 41, and the lower the score, the better the state.